CLINICAL TRIAL: NCT04648514
Title: Radiographic Evaluation of Bone Height Gain With Dental Implant Placed Simultaneously With Closed Sinus Lifting Using Hydraulic Lift Technique Versus Summers' Osteotome Technique in Posterior Edentulous Maxilla (Randomized Clinical Trial)
Brief Title: Radiographic Evaluation of Bone Height Gain With Dental Implant Placed Simultaneously With Closed Sinus Lifting Using Hydraulic Lift Technique Versus Summers' Osteotome Technique in Posterior Edentulous Maxilla (RCT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohammad, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7920
Record Dates: First submitted 2020-11-15; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Evaluations, Diagnostic Self

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using of bone osteotomes for closed sinus lifting (Active Comparator): Using of summers' osteotome technique by bone osteotomes for closed sinus lifting then evaluation the amount of bone height gain will be done radiographically (by panorama and CBCT) after implant placement in posterior edentulous maxilla .
  Interventions: Procedure: Using of hydraulic lifter device for closed sinus lifting
- Patient satisfaction evaluation after using bone osteotomes (Active Comparator): Evaluation of patient satisfaction numerically will be done after using summers' osteotome technique by bone osteotomes for closed sinus lifting in posterior edentulous maxilla
  Interventions: Behavioral: patient satisfaction evaluation after using hydraulic lifter device

INTERVENTIONS:
Procedure: Using of hydraulic lifter device for closed sinus lifting — Using of recent closed minimally invasive technique (hydraulic left technique) by hydraulic lifter device for closed sinus lifting then evaluation of the amount of bone height gain will be done radiographically (by panorama and CBCT) after implant placement for patients with posterior edentulous maxilla .
  Arms: Using of bone osteotomes for closed sinus lifting
Behavioral: patient satisfaction evaluation after using hydraulic lifter device — Evaluation of patient satisfaction numerically will be done after using hydraulic lift technique by hydraulic lifter device for closed sinus lifting in posterior edentulous maxilla
  Arms: Patient satisfaction evaluation after using bone osteotomes

SUMMARY:
Radiographic evaluation of bone height gain with dental implant placed simultaneously with closed sinus lifting using hydraulic lift technique versus summers' osteotome technique in posterior edentulous maxilla (RCT)

DETAILED DESCRIPTION:
Evaluation will be done on the amount of bone height gain radiographically (using both panorama and CBCT) after placement of the dental implant simultaneously with closed sinus lifting using hydraulic lift technique versus summers' osteotome technique in patients with posterior edentulous maxilla (Randomized Clinical Trial)

ELIGIBILITY:
Inclusion Criteria:

* Edentulous patients in the maxillary posterior region .
* Patients in need to fixed restorations in posterior region .
* Patients with a healthy systemic conditions.(Apparently medically free)
* Patients with adequate inter-arch space for placement of the prosthetic part of the implant .
* Patients who had approximately 5-8 mm of available bone height between crest of bone and floor of sinus
* Both sexes.
* Patients with Good oral hygiene
* Patients more than 20 years old
* Cooperative and motivated patients

Exclusion Criteria:

* Patients with local pathological defects related to posterior maxilla .
* Heavy smokers.
* Abnormal habits that may alter results such as alcoholism or parafuctional habits .
* Patients with systemic diseases that may affect normal healing.
* Patients with psychiatric problem
* Patients with history of recent radiation therapy to the head and neck area .
* Patients with aggressive periodontitis .

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Amount of bone height change | 6 months
  Evaluation of the amount of bone height change radiographically after closed sinus lift simultaneously with implant placement using hydraulic lift technique versus summers' osteotome technique in posterior edentulous maxilla

SECONDARY OUTCOMES:
Patient satisfaction numerical questionnaire | 6 months
  Evaluation of patient satisfaction by using specific numerical questionnaire which depends on numerical scale after closed sinus lifting procedure with implant placement using hydraulic lift technique versus summers' osteotome technique in posterior edentulous maxilla .
  The patient satisfaction numerical questionnaire include several questions to the patient and the patient will put a circle sign on the mark at which he or she feels to represent the answer .
  The numerical scale is from 1 to 5 for each question (with total of 20 questions) :
  1. represents strongly disagree
  2. represents disagree
  3. represents neither agree or disagree
  4. represents agree
  5. represents strongly agree
  The final score is out of 100 so, more higher scores represents more patient satisfaction and so, better outcome and less scores represents less patient satisfaction and so, worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Abdelghany, PHD, Study Director — Assoc.professor of oral and maxillofacial surgery
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No